CLINICAL TRIAL: NCT00752297
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Two-Arm, Single-Dose Pivotal Trial to Demonstrate the Safety and Efficacy of PurTox® for the Treatment of Glabellar Rhytides ("Frown Lines")
Brief Title: Safety and Efficacy Study of PurTox® Botulinum Toxin Type A to Treat Frown Lines Between the Eyebrows
Acronym: PT-03a
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-03a
Record Dates: First submitted 2008-09-10; First posted 2008-09-15 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Glabellar Rhytides
Keywords: Botulinum Toxin Type A; Botulinum Toxin; Glabellar Rhytides; Rhytides; Frown Lines; Neuromuscular Agents; Neurotoxin; Forehead; Eyebrow; Wrinkle
MeSH Terms: interventions — Sodium Chloride; Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mentor Purified Toxin Botulinum Toxin Type A
  Interventions: Drug: Mentor Purified Toxin
- 2 (Placebo Comparator): Preservative-free Saline
  Interventions: Drug: Preservative-free Saline

INTERVENTIONS:
Drug: Preservative-free Saline — Subjects will receive five 0.1 mL intramuscular injections at the Day 0 Treatment Visit: two in each corrugator and one in the procerus muscle. The total treatment dose (sum of the five injections) to be administered will be 0.5 mL of the placebo (preservative-free saline).
  Other Names: Saline
  Arms: 2
Drug: Mentor Purified Toxin — All subjects will receive five 0.1 mL intramuscular injections (two in each corrugator and one in the procerus muscle) at each Treatment Visit. The total treatment dose (sum of the five injections) to be administered will be 30 U of PurTox. Subjects will have many Treatment Visits throughout the course of the three-year study.
  Other Names: Arms: 1; Other Names:; Mentor Purified Toxin Botulinum Toxin Type A; Botulinum Toxin Type A; Botulinum Toxin
  Arms: 1

SUMMARY:
The overall purpose of this study is to evaluate the safety and effectiveness of an intramuscular dose of Mentor Purified Toxin for the reduction of frown lines, compared with placebo.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, randomized, double-blind, placebo-controlled, two-arm, single-dose study to evaluate the safety and efficacy of Mentor Purified Toxin for the treatment of glabellar rhytides. Approximately 400 subjects will be enrolled in the study. The subjects will be randomized 3:1 (300 Mentor Purified Toxin: 100 placebo) to receive either intramuscular injections of 30 U of Mentor Purified Toxin or placebo (preservative-free saline).

Injected subjects will be observed for 180 days of post treatment follow-up. Follow-up clinic visits are scheduled for post treatment days 3, 7, 14, 30, 60, 90, 120, 150, and 180.

The study will be conducted at up to ten clinical sites. Safety, tolerability, clinical efficacy, onset and duration of effect will be studied during the study

The effectiveness of Mentor Purified Toxin will be determined by the degree of frown line reduction, during maximum forced frown and at rest (neutral expression):

* as assessed live by the study doctor,
* as assessed live by the subject, and
* as assessed by an independent reviewer based on subject photographs

Frown lines are graded on level of severity based on this scale:

Severity

* Minimal (0)
* Mild (1)
* Moderate (2)
* Severe (3)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are 18 years of age or older (subjects should have an interest in the effacement of glabellar rhytides) with or without previous botulinum Toxin Type A exposure;
2. In good physical and mental health as determined by the investigator based on medical history, physical examination, and/or clinical laboratory tests;
3. Noticeable presence of the glabellar rhytides for a period of 6 months or longer;
4. Score at least a 2 (moderate severity) at baseline screening on the investigator's and subject's assessments (reference photographs provided) at forced frown; and
5. Capable of understanding and complying with the protocol and must have signed the informed consent document prior to performance of any study-related procedures.

Exclusion Criteria:

1. History of psychiatric problems that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
2. History of autoimmune disease, that, in the opinion of the investigator, might interfere with subject outcomes (e.g., osteoarthritis is not considered an exclusion criteria; however, subjects with dermatomyositis are not permitted to participate in this study);
3. History or presence of clinically significant cardiovascular, respiratory, hepatic/biliary, renal, gastrointestinal, endocrinological, or neurological disorders constituting a possible risk factor that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
4. Inability to substantially efface glabellar lines by manually spreading skin apart;
5. Eyelid ptosis;
6. Myasthenia gravis (from medical history or diseases of neurotransmission);
7. Current history of facial nerve paralysis;
8. Concurrent dermatologic disease of the face in the glabellar area that is deemed by the investigator to make the subject an inappropriate candidate for the study;
9. Recent flu-like syndrome that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
10. Neuromuscular disorder that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
11. Active multisystems disease that, in the investigator's opinion, might influence the outcome measures or the safety of the subject;
12. Has any condition(s) that in the investigator's opinion would a) warrant exclusion from the study, or b) prevent the subject from completing the study;
13. Currently receiving aminoglycoside antibiotic therapy, curare-like drugs, quinidine, succinylcholine, polymyxins, anticholinesterases, magnesium sulfate, or lincosamides;
14. Has taken any investigational drug during the 30 days prior to screening visit;
15. Have had Botulinum Toxin treatments to the glabellar and/or forehead area during the 6 months prior to screening visit;
16. Have had dermal filler treatment to glabellar area during the 6 months prior to screening visit;
17. Female subjects who are pregnant or lactating. (Female subjects of childbearing potential must have negative urine pregnancy test results prior to enrollment into the study. Such subjects, including peri-menopausal women who have had a menstrual period within one year, must use appropriate birth control (see protocol/informed consent for description)
18. Unwilling or unable to comply with the protocol or to cooperate fully with the investigator and site personnel; and
19. Unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent document is available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Degree of glabellar rhytide reduction assessed by the investigator and the subject at maximum frown as a single composite effectiveness endpoint. | Day 30 post-injection
Measurement of the incidences of treatment-emergent adverse events, serious treatment-emergent adverse events, treatment-emergent laboratory abnormalities, and vital signs. | Throughout

SECONDARY OUTCOMES:
Degree of glabellar rhytide reduction assessed by the investigator and the subject at maximum frown. | Days 3, 7 and 30 post-injection
Degree of glabellar rhytide reduction assessed by the investigator and the subject at rest. | Day 30 Post-injection
Degree of glabellar rhytide reduction assessed by independent reviewers based on photographs of the subject's glabellar lines at maximum frown. | Baseline and Day 30 post-injection
Explore the global satisfaction of the subject with the treatment. | Day 30 post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Corey Maas, MD, Study Director
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States